CLINICAL TRIAL: NCT04187209
Title: Evaluation of the Use of the Atalante System in Patients Presenting a Non-traumatic Hemiplegia in Acute-subacute Phase (15 Days to 6 Months).
Acronym: SPIRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPIRIT
Record Dates: First submitted 2019-11-15; First posted 2019-12-05 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Stroke, Acute; Stroke, Subacute; Robotics
Keywords: Stroke; Acute Stroke; Subacute Stroke; Robotics; Physiotherapy; Rehabilitation; Powered exoskeleton; Walking; Exercises; Ambulation
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-traumatic hemiplegia in post stroke acute subacute phase (Other)
  Interventions: Device: Use of the Atalante exoskeleton

INTERVENTIONS:
Device: Use of the Atalante exoskeleton — A session includes a stand-up, walks over a distance of 10 meters, exercises with or without the assistance of the exoskeleton, U-turns and a sitting.

SUMMARY:
The SPIRIT study is interventional, national, prospective, open, multicentric each patient being his/her own control.

It is conducted to assess the safety and performance of the Atalante exoskeleton system in patients presenting a non-traumatic acute-subacute hemiplegia. The primary endpoint is defined by the patient's ability to perform the 10 MWT with the Atalante system.

The study will include at least 12 patients and takes place in three french rehabilitation centers.

ELIGIBILITY:
Inclusion Criteria:

* Patient with non-traumatic vascular hemiplegia in acute subacute phase (15 days to 6 months) hospitalized in rehabilitation center,
* Patients presenting a FAC score of 0, 1 or 2,
* Patient with ischemic or hemorrhagic stroke of which etiological evaluation is complete,
* Adult patient ≥18 years old,
* Patient able to verticalize on a daily basis and having a stabilized blood pressure,
* Patient with stable medical condition at the time of inclusion in the study (absence of infectious and cardiorespiratory events),
* Patient's height is at least 1m55,
* Lengths of patient's lower limb are in the following intervals:

  * Thigh (distance gluteus maximus - patella): 56.8 and 64.8 cm,
  * Distance between the ground and the joint space of the knee (to be measured while wearing the shoes the patient intends to wear with Atalante):

    * 45.7-60.7 cm for patient with an ankle dorsiflexion ≥ 16°
    * 45.7-57.7 cm for patient with an ankle dorsiflexion > 13° et < 16°
    * 45.7-56.7 cm for patient with an ankle dorsiflexion > 10° et ≤ 13°
    * 45.7-55.7 cm for patient with an ankle dorsiflexion ≥ 0° et ≤ 10°
  * Intertrochanteric distance lower or equal to 46.0 cm when seated,
* Maximum weight: 90 kg,
* Patient able to read and write French and who have signed an informed consent form.

Exclusion Criteria:

* Ranges of motion below:

  * Hip: 90° flexion, 5° extension, 17° abduction, 10° adduction, 10° medial rotation, 20° lateral rotation
  * Knee: 5° extension, 110° flexion
  * Ankle: 0° dorsiflexion, 9° plantar flexion, 18° inversion and eversion
* Patient whose joint centers cannot be aligned Atalante's system,
* Severe spasticity (greater than 3 on the modified Ashworth scale) of the adductor muscles, hamstrings, quadriceps and triceps surae
* Pregnant or lactating women,
* Medical history of osteoporotic fracture and/or disease or treatment responsible for a secondary osteoporosis,
* Patient with a cardiac contraindication to physical exertion,
* Evolutive intercurrent disease: venous thrombosis, hypotension,
* Patient unable to deliver his/her consent,
* Patient under legal protection,
* Patient participating at the same time in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the use of the Atalante system in patients with non-traumatic acute-subacute hemiplegia over several sessions with a 10 meter Walk Test. This test will show the incidence of test success and emergence of adverse events. | At study mid-term, 6 days in average
  Defined by the patient's ability to perform the 10mWT with the Atalante system.
Evaluate the use of the Atalante system in patients with non-traumatic acute-subacute hemiplegia over several sessions with a 10 meter Walk Test. This test will show the incidence of test success and emergence of adverse events. | At study mid-term, 7 days in average
  Defined by the patient's ability to perform the 10mWT with the Atalante system
Evaluate the use of the Atalante system in patients with non-traumatic acute-subacute hemiplegia over several sessions with a 10 meter Walk Test. This test will show the incidence of test success and emergence of adverse events. | At study mid-term, 8 days in average
  Defined by the patient's ability to perform the 10mWT with the Atalante system
Evaluate the use of the Atalante system in patients with non-traumatic acute-subacute hemiplegia over several sessions with a 10 meter Walk Test. This test will show the incidence of test success and emergence of adverse events. | At study completion, 9 days in average
  Defined by the patient's ability to perform the 10mWT with the Atalante system
Evaluate the use of the Atalante system in patients with non-traumatic acute-subacute hemiplegia over several sessions with a 10 meter Walk Test. This test will show the incidence of test success and emergence of adverse events. | At study completion, 10 days in average
  Defined by the patient's ability to perform the 10mWT with the Atalante system

SECONDARY OUTCOMES:
Evaluate the patient's ambulatory ability without the Atalante exoskeleton with the Functional Ambulation Classification (FAC). | At baseline, day 0 and at study completion, up to 10 days
  Evaluation of the walk performance with the FAC classification.
  0: Nonfunctional ambulation
  1. Ambulator-Dependent for Physical Assistance Level II
  2. Ambulator-Dependent for Physical Assistance Level I
  3. Ambulator-Dependent for Supervision
  4. Ambulator-Independent Level Surfaces only
  5. Ambulator-Independent
Evaluate the settings of the walking parameters of the exoskeleton deemed most efficient by the patient (step length, cadence) | Day 2 until study mid term, day 5
  During sessions 2 to 5, the physiotherapist will vary the step length and cadence of the exoskeleton's walk.
  Each parameter will be tested over a distance of 10 meters. Perceived exertion and perceived safety will be assessed by the patient using a Likert Scale. Physiotherapist satisfaction (evaluated on a Likert Scale) will be assessed at the end of the test.
  Likert scale :
  1. "Strongly disagree"
  2. "Disagree"
  3. "Neither agree or disagree"
  4. "Agree"
  5. "Strongly agree"
Evaluate the assistive control settings | Day 2, day 4
  The test of dynamic assistance is performed in WALK mode. The patient starts by leaning the right side (or left side). Then, as soon as the user presses WALK button, a first step is triggered by the exoskeleton. Next steps are more or less assisted depending on the level of assistance chosen by the physiotherapist (100% of assistance equals 0% effort of the patient, Atalante performs the movement instead of the patient). The patient must initiate each step by pushing on the opposite leg and making a pelvic rotation towards the forward foot.
  Values of tested assistance levels assessed will be collected as perceived exertion, perceived safety and physiotherapist satisfaction (evaluated on a Likert Scale).
  Likert scale :
  1. "strongly disagree"
  2. "disagree"
  3. "neither agree or disagree"
  4. "agree"
  5. "strongly agree",
Evaluate the patient's ability to perform weight transfer on the hemiplegic side or the healthy side | Day 2, day 4
  Success/ Failure to the exercise: transfer of weight to the right or left side until the sound signal is triggered
Evaluate the patient's ability to perform a semi-squat | Day 3, day 5
  Success/ Failure to the exercise: perform a semi-squat
Evaluate the level of assistance needed by the patient from the healthcare staff to perform tests | Throughout study completion, an average of 10 days
  The therapist will record the level(s) of assistance needed to perform each test and detail the moment on which assistance was needed during the test. The level of assistance will be determined with the number of times the therapist will have helped the patient during the tests, as well as the type of assistance he/she will have provided.
  The physiotherapist will select on a scale the level of assistance he/she provided during the test:
  * None (0% of assistance)
  * Minimal (0-25% assistance)
  * Moderate (25-50% assistance)
  * High (50-75% assistance)
  * Maximum (75-100% assistance).
Evaluate the time needed for the patient to don and doff | At study completion, day 10
  Collection of data regarding the time needed for patient to donning and doff
Evaluate the patient's physical and cognitive conditions using the Berg Balance Scale | At baseline, day 0 and at study completion, up to 10 days
  The Berg Balance Scale (BBS) is a 14-item objective measure that assesses static balance and risk of fall in adult. In this 14-item scale, patient must maintain positions and complete moving tasks of varying difficulty. In most items, patient must maintain a given position for a specified time. Patient receives a score from 0-4 on his/her ability to meet these balance dimensions:
  * 0-20 on the BBS represents balance impairment;
  * 21-40 on the BBS represents acceptable balance;
  * 41-56 on the BBS represents good balance.
  This measure will be performed during sessions 0 and 10 in order to assess a potential variation
Evaluate the patient's physical and cognitive conditions | At baseline, day 0
  Evaluation of the level of aphasia by the aphasia severity rating scale from the Boston Diagnostic Aphasia Examination.
  The degree of aphasia will be evaluated using the aphasia severity rating scale from the Boston diagnostic Aphasia Examination (BDAE). BDAE is designed to diagnose aphasia and related disorders. This test evaluates the various conceptual modalities (auditory, visual and gestural), the processing functions (comprehension, analysis, problem solving) and the response modalities (writing, articulation and manipulation).
  The aphasia severity rating scale from the BDAE will be done at baseline in order to describe the population participating in the study.
Evaluate the level of effort perceived during each test by using the Borg scale | Throughout study completion, an average of 10 days
  Rating of perceived exertion (RPE) will be used to assess the effort perceived by patient at each session. RPE is a widely used and reliable indicator to monitor and guide exercise intensity. The scale allows individuals to subjectively rate their level of exertion during exercise or exercise testing.
  The revised category-ratio scale (0 to 10 scale) is used:
  0 Null
  1. Very easy
  2. Somewhat easy-
  3. Moderate
  4. Somewhat hard
  5. Hard
  7 Very hard 8 9 10 Very, very hard
Evaluate the level of security perceived during each test by using a 5-level Likert scale | Throughout study completion, an average of 10 days
  Perceived safety during tests will be assessed by each patient using a 5-point Likert scale format ranging from 5)"strongly agree", 4)"agree", 3)"neither agree or disagree", 2)"disagree" and 1)"strongly disagree".
  The range of Likert scale captures the intensity of his/her feeling for a given item.
Evaluate the level of anxiety of patient related to the use of the exoskeleton | At study start, day 1 and at study completion, up to 10 days
  Collection of the patient's level of anxiety assessed by a 5-level Likert scale:
  1. "strongly disagree"
  2. "disagree"
  3. "neither agree or disagree",
  4. "agree",
  5. "strongly agree",
Evaluate the emergence of musculoskeletal disorders in the therapist | At baseline, day 0 and at study completion, up to 10 days
  Evaluation of musculoskeletal disorders developed by healthcare professionals in the use of exoskeleton with a Nordic style questionnaire.
  The Nordic Musculoskeletal Questionnaire (NMQ) is a 2-section questionnaire. The aim was to develop and test a standardized questionnaire methodology allowing comparison of low back, neck, shoulder and general complaints.
  The NMQ can be used as a questionnaire or as a structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kerdraon, Dr, Principal Investigator — Centre mutualiste de Rééducation et de Réadaptation de Kerpape; Jean-Gabriel Prévinaire, Dr, Principal Investigator — Centre Jacques Calvé - Fondation Hopale de Berck-sur-Mer; Soultana Tatsidou, Dr, Principal Investigator — Centre de Médecine Physique et de Réadaptation de Pionsat
Locations (3):
- France (3):
  - Centre Jacques Calvé - Fondation Hopale, Berck
  - Centre de Médecine Physique et de Réadaptation de Pionsat, Pionsat
  - Centre mutualiste de Rééducation et de Réadaptation de Kerpape, Ploemeur